CLINICAL TRIAL: NCT01199016
Title: "a Phase 4, Postmarketing Study Evaluating The Impact Of Prevnar 13 (Trademark)(13-valent Pneumococcal Conjugate Vaccine; 13vpnc) In Reducing Acute Otitis Media And Nasopharyngeal Colonization Caused By Streptococcus Pneumoniae In Healthy Children
Brief Title: Effect of Prevnar 13 on Ear Infections in Children
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 6096A1-4010; B1851018 (Other: Alias Study Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2016-12

CONDITIONS: Otitis Media
Keywords: Acute otitis media; Prevnar 13; Streptococcus pneumoniae; nasopharyngeal colonization.
MeSH Terms: conditions — Otitis Media | interventions — Tympanocentesis; Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle Ear Fluid for microbiologic analysis Nose and throat swab for microbiologic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Tympanocentesis; Procedure: Nose/throat swab; Biological: Observational

INTERVENTIONS:
Procedure: Tympanocentesis — To be performed as needed on children presenting with acute otitis media
Procedure: Nose/throat swab — To be performed at every study visit
Biological: Observational — Observational Study Only

SUMMARY:
Prevnar (7 valent pneumococcal conjugate vaccine [7vPnC]) has been shown to be effective against ear infections in children. Prevnar 13 is a new vaccine that is similar to Prevnar. It is expected that the effectiveness of Prevnar 13 against ear infections in children will be similar to that observed following Prevnar. Pfizer has committed to conduct a postmarketing study of the impact of Prevnar 13 in reducing ear infections among children.

DETAILED DESCRIPTION:
Infants who have completed the Prevnar 13 infant vaccination series who provide consent and fit the study inclusion criteria to participate in the study will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Subject has received full (3-dose) infant series of Prevnar 13

Exclusion Criteria:

* Prior vaccination with any 7vPnC.
* Prior vaccination with 23-valent pneumococcal polysaccharide vaccine (23vPS).
* Any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in the study.

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy children aged approximately 6 to 36 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2010-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Penfield Pediatrics, Penfield, New York
  - Long Pond Pediatrics, Rochester, New York
  - Legacy Pediatrics, Rochester, New York
  - Lewis Pediatrics, Rochester, New York
  - Pathway Pediatrics, Rochester, New York
  - Sunrise Pediatrics, Rochester, New York
  - Westfall Pediatrics, Rochester, New York

REFERENCES:
- [Derived] Pichichero M, Kaur R, Scott DA, Gruber WC, Trammel J, Almudevar A, Center KJ. Effectiveness of 13-valent pneumococcal conjugate vaccination for protection against acute otitis media caused by Streptococcus pneumoniae in healthy young children: a prospective observational study. Lancet Child Adolesc Health. 2018 Aug;2(8):561-568. doi: 10.1016/S2352-4642(18)30168-8. Epub 2018 Jun 19. PMID 30119715
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-4010&StudyName=Effect%20of%20Prevnar%2013%20on%20Ear%20Infections%20in%20Children

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevnar 13: Participants who were 6 to 12 months of age and had completed immunization schedule of the Prevnar 13 infant series or participants who were up to 30 months of age and met the criteria for recurrent acute otitis media (AOM) were enrolled. Recurrent AOM was defined as greater than or equal to (>=)3 distinct episodes in a 6-month period or >=4 distinct episodes in a 12-month period. Participants who were diagnosed with AOM, underwent both nasopharyngeal/oropharyngeal (NP/OP) swab and diagnostic tympanocentesis (or collection of MEF via swab if tympanocentesis could not be performed).
Period: Overall Study
Arm/Group | Prevnar 13
Started | 239
Treated | 236
Completed | 162
Not Completed | 77
Not completed — No longer meets eligibility criteria | 4
Not completed — Entrance criteria | 5
Not completed — Protocol Violation | 9
Not completed — Other | 13
Not completed — Withdrawal by Subject | 21
Not completed — Lost to Follow-up | 25

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had at least one dose of study drug and had undergone at least 1 of the study procedures.
Arm/Group | Prevnar 13
Number analyzed (Participants) | 236
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.4 (2.61)
Gender [Count of Participants; unit: Participants]
  Female | 115
  Male | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Middle Ear Fluid (MEF) Samples With Positive Results for Streptococcus Pneumoniae Serotypes 1, 3, 5, 6A, 7F, or 19A in Participants With Acute Otitis Media (AOM)
Description: MEF samples were obtained from participants who presented with an episode of AOM as defined by clinical criteria. Total percentage of MEF samples that were tested positive for any of the 6 additional serotypes included in Prevnar 13 (1, 3, 5, 6A, 7F, or 19A) have been reported.
Time Frame: Baseline up to Month 36
Population: MEF AOM population included all participants with at least 1 MEF sample from an episode of AOM. In this analysis, 'Number of MEF samples analyzed' indicates those samples that tested positive for Streptococcus pneumoniae serotypes 1, 3, 5, 6A, 7F, or 19A.
Measure: Number; unit: percentage of MEF samples
Units Other Than Participants: MEF Samples
Arm/Group | Prevnar 13
Number analyzed (Participants) | 90
Number analyzed (MEF Samples) | 53
percentage of MEF samples | 7.5

2. Other Pre Specified Outcome: Percentage of Nasopharyngeal/Oropharyngeal (NP/OP) Samples With Positive Results for Streptococcus Pneumoniae Serotypes 1, 3, 5, 6A, 7F, or 19A in Healthy Participants
Description: Total percentage of NP/OP samples that were tested positive for any of the 6 additional serotypes included in Prevnar 13 (1, 3, 5, 6A, 7F, or 19A) have been reported. NP/OP samples were collected from participants at all healthy visits as well as AOM visits.
Time Frame: Baseline up to Month 36
Population: NP/OP healthy population included all participants with an NP/OP swab collection at a healthy visit. In this analysis, 'Number of NP/OP samples analyzed' indicates those samples that tested positive for Streptococcus pneumoniae serotypes 1, 3, 5, 6A, 7F, or 19A.
Measure: Number; unit: percentage of NP/OP samples
Units Other Than Participants: NP/OP Samples
Arm/Group | Prevnar 13
Number analyzed (Participants) | 228
Number analyzed (NP/OP Samples) | 383
percentage of NP/OP samples | 6.0

3. Other Pre Specified Outcome: Percentage of Middle Ear Fluid (MEF) Samples With Positive Results for Streptococcus Pneumoniae Serotypes Other Than 1, 3, 5, 6A, 7F, or 19A in Participants With Acute Otitis Media (AOM)
Description: MEF samples were obtained from participants who presented with an episode of AOM as defined by clinical criteria. Total percentage of MEF samples that were tested positive for Streptococcus pneumoniae serotypes other than those included in Prevnar 13 (1, 3, 5, 6A, 7F, or 19A) have been reported.
Time Frame: Baseline up to Month 36
Population: MEF AOM population included all participants with at least 1 MEF sample from an episode of AOM. In this analysis, 'Number of MEF samples analyzed' indicates those samples that tested positive for Streptococcus pneumoniae.
Measure: Number; unit: percentage of MEF samples
Units Other Than Participants: MEF Samples
Arm/Group | Prevnar 13
Number analyzed (Participants) | 90
Number analyzed (MEF Samples) | 53
percentage of MEF samples | 92.5

4. Other Pre Specified Outcome: Percentage of Nasopharyngeal/Oropharyngeal (NP/OP) Samples With Positive Results for Streptococcus Pneumoniae Serotypes Other Than 1, 3, 5, 6A, 7F, or 19A in Healthy Participants
Description: Total percentage of MEF samples that were tested positive for Streptococcus pneumoniae serotypes other than those included in Prevnar 13 (1, 3, 5, 6A, 7F, or 19A) have been reported. NP/OP samples were collected from participants at all healthy visits as well as AOM visits.
Time Frame: Baseline up to Month 36
Population: NP/OP healthy population included all participants with an NP/OP swab collection at a healthy visit. In this analysis, 'Number of NP/OP samples analyzed' indicates those samples that tested positive for Streptococcus pneumoniae.
Measure: Number; unit: percentage of NP/OP samples
Units Other Than Participants: NP/OP Samples
Arm/Group | Prevnar 13
Number analyzed (Participants) | 228
Number analyzed (NP/OP Samples) | 383
percentage of NP/OP samples | 94.0

ADVERSE EVENTS:
Description: Only protocol-related adverse events (AEs) or research-related injury (RRIs) were planned to be collected.
Arm/Group | Prevnar 13
Serious Adverse Events (participants affected / at risk) | 0/239
Other Adverse Events (participants affected / at risk) | 0/239

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.